CLINICAL TRIAL: NCT03758950
Title: Inhaled Mometasone to Promote Reduction in Vasoocclusive Events 2
Acronym: IMPROVE2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jeffrey Glassberg (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Jeffrey Glassberg, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 17-1936; R01HL142671 (NIH)
Record Dates: First submitted 2018-11-28; First posted 2018-11-29 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell; Inhaled Steroids
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Once daily inhaled placebo
  Interventions: Drug: Placebo
- Mometasone (Active Comparator): Inhaled Mometasone Furoate 220 mcg DPI
  Interventions: Drug: Mometasone

INTERVENTIONS:
Drug: Placebo — Once daily inhaled placebo for 48 weeks
  Arms: Placebo
Drug: Mometasone — Inhaled Mometasone for 48 weeks (with 4-week washout at study completion)
  Other Names: Inhaled Mometasone
  Arms: Mometasone

SUMMARY:
The study team proposes a triple-blind, placebo-controlled, phase II clinical trial of once-daily inhaled mometasone for 48 weeks (with 4-week washout at study completion) in individuals with Sickle Cell Disease (SCD) who report episodic cough or wheeze (ECW) but do not have asthma. Patients will be recruited from and followed in SCD clinics at participating sites. The primary endpoint will be a reduction in sVCAM level of 20% or more in comparison to placebo.

DETAILED DESCRIPTION:
Dose rationale: Mometasone furoate 220mcg dry powder inhalation is a low-moderate ICS dose that can be given once daily. Higher doses can have systemic effects and systemic glucocorticoids can precipitate rebound SCD pain when discontinued.

Adaptive, covariate-balanced randomization: While the sample size of the study will be fixed at 80 participants, instead of standard blocked or stratified randomization, the study team will use adaptive covariate-balanced randomization to minimize imbalance of important covariates. This will reduce the need to use multivariable techniques (which perform poorly in small samples) to adjust post hoc for differences between treatment groups. Covariates will include age, use of hydroxyurea, previous rate of Emergency Department (ED) utilization for SCD pain, and recruitment site.

Follow up Schedule: There will be in-person visits every 8 weeks. In addition, a blinded research coordinator will contact participants by phone at 2-weeks and 4-weeks after enrollment and 4-weeks after each in-person follow up to encourage protocol adherence and collect data about adverse events and healthcare utilization.

Post-protocol observation period: The study will be complete at 48 weeks. A final follow up visit will occur at 52 weeks (4-weeks after study protocol completed) to collect pain diary and adverse event data and to identify the proportion of the ICS group who want to continue ICS. In the event that individuals wish to continue ICS, the PI will contact the participant's treating physician to discuss.

Data elements: A wide range of clinical and translational data will be collected during the study. Baseline data will include demographic and clinical variables regarding SCD severity, previous complications and respiratory surveys. Blood will be collected for standard-of-care labs and analysis of serum inflammatory cytokines. Pulmonary function testing including spirometry and Exhaled Nitric Oxide (eNO) will be performed. Health related quality of life will be collected via ASCQ-Me survey. Patients will also be followed with follow-up phone calls and prospective chart review for one year to identify hospital visits and other SCD complications.

Procedures for collection of clinical and laboratory data: Data collection and management: Case report forms are provided as an appendix. Data will be entered into a REDCap database, which will be monitored by the Data Coordinating Team (DCT) (led by Co-I Gelijns) for completion and timeliness.

ELIGIBILITY:
Inclusion Criteria:

* Participants age 18 and older with severe SCD phenotypes (Hb SS and Sβthalassemia0):
* Do not have asthma (see exclusion criteria)
* Not currently having a painful crisis (as defined by validated pain diary questions)
* Do not have acute respiratory symptoms
* Report of recent ECW (answers "Yes" to any question in Box 1)
* Participant is already medically optimized (i.e. already on maximum dose hydroxyurea unless contraindicated and not undergoing medication titration).

Exclusion Criteria:

* Participant screens positive for possible undiagnosed asthma (Box 2)
* Pregnant or planning to become pregnant
* > 15 ED visits for SCD pain over the previous 12 months (due to concern for multi-factorial pain that may be less responsive to SCD therapies)
* Have been discharged from the hospital within the previous 7 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Soluble Vascular Cell Adhesion Molecule (sVCAM) level | Baseline and one year
  Change in sVCAM level at one year compared to baseline. sVCAM is a biomarker used as a surrogate for red blood cell (RBC) adhesivity and overall disease severity in SCD.

SECONDARY OUTCOMES:
Reticulocyte Count level | Baseline and one year
  Change in Reticulocyte Count level at one year compared to baseline. Reticulocyte count is a secondary measure of hemolysis. In SCD, it is more reflective of hemolytic burden than any other clinically available laboratory test.
Plasma Free Hemoglobin level | Baseline and one year
  Change in Free Hemoglobin level at one year compared to baseline. Free hemoglobin is a direct measure of hemolysis. It is more reflective of hemolytic burden than reticulocyte count but it is not available for clinical use.
LDH level | Baseline and one year
  Change in LDH level at one year compared to baseline. LDH is a marker of hemolysis
Bilirubin (Direct and Indirect) level | Baseline and one year
  Change in Bilirubin level at one year compared to baseline. Bilirubin measure of hemolysis
Hemoglobin level | Baseline and one year
  Change in Hemoglobin level at one year compared to baseline. Hemoglobin is a clinical lab test
Leukocyte Count level | Baseline and one year
  Change in Leukocyte level at one year compared to baseline. Leukocyte is a clinical lab test
Platelet Count level | Baseline and one year
  Change in Platelet count level at one year compared to baseline. Platelet count is a clinical lab test
Exhaled Nitric Oxide | Baseline and one year
  Change in eNO level at one year as compared to baseline. Nitric oxide is a marker of eosinophilic pulmonary inflammation
Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-Me) survey | Baseline and one year
  ASCQ-Me is a patient-reported outcome measurement system that evaluates and monitors the physical, mental, and social well-being of adults with sickle cell disease (SCD). ASCQ-Me uses a T-score metric in which 50 is the mean of the reference population and 10 is the standard deviation (SD) of that population.
Medication Adherence Self-Report Scale for Asthma (MARS-A) | At one year
  MARS-A is a 10-item, self-reported measure of adherence
Brain Natriuretic Peptide | Baseline and one year
  Change in brain natriuretic peptide at one year compared to baseline. Brain natriuretic peptide is a measure of atrial stretch.
Spirometry | Baseline and one year
  Change in spirometry at one year compared to baseline. Spirometry is the measure of airflow and lung function.
Pain Score | Up to one year
  Pain score on a zero to ten scale reflects "yesterday's worst pain".
Number of ED Visits for SCD Pain | One year
  Measure of morbidity and healthcare utilization
Number Hospitalizations for SCD Pain | One year
  Measure of morbidity and healthcare utilization
Number of Observation Unit Admission for SCD Pain | One year
  Measure of morbidity and healthcare utilization
Number of Overnight Stays for SCD Pain | One year
  Measure of morbidity and healthcare utilization
Number of Outpatient Infusion Visits for SCD Pain | One year
  Measure of morbidity and healthcare utilization
Number of Pneumonia Episodes | One year
  Measure of morbidity and healthcare utilization
Number of ICU Admissions | One year
  Measure of morbidity and healthcare utilization
Number of Deaths | One year
  Measure of disease severity
O-Link Inflammation Panel Serum | Baseline and one year
  Change in O-Link Inflammation Panel Serum at one year compared to baseline. A 92 analyte panel of key molecules involved in inflammation
O-Link Inflammation Panel Sputum | Baseline and one year
  Change in O-Link Inflammation Panel Sputum at one year compared to baseline. Inflammation panel performed on sputum supernatant will be a measure of pulmonary inflammatory signatures
Multiplex Cytokine Panel Serum | Baseline and one year
  Change in Multiplex Cytokine Panel Serum at one year compared to baseline. Key inflammatory mediators including interleukins, selectins, interferon and TNF.
Sputum frequency of activated monocytes CyTOF | Baseline and one year
  Change in Sputum frequency of activated monocytes CyTOF at one year compared to baseline. Measure of pulmonary inflammation
Sputum Frequency of Aged Neutrophils CyTOF | Baseline and one year
  Change in Sputum Frequency of Aged Neutrophils CyTOF at one year compared to baseline. Measure of pulmonary inflammation
Sputum Immune Cell Subpopulations CyTOF | Baseline and one year
  Change in Sputum Immune Cell Subpopulations CyTOF at one year compared to baseline. Frequencies of all immune subpopulations will be calculated to identify pulmonary inflammation signatures.
Sputum Immune Cell Subpopulations CyTOF | Baseline and one year
  Change in Sputum Immune Cell Subpopulations CyTOF at one year compared to baseline. Measure of pulmonary inflammation
Whole Blood Frequency of Aged Neutrophils CyTOF | Baseline and one year
  Change in Whole Blood Frequency of Aged Neutrophils CyTOF at one year compared to baseline. Measure of pulmonary inflammation
Whole Blood Immune Cell Subpopulations CyTOF | Baseline and one year
  Change in Whole Blood Immune Cell Subpopulations CyTOF at one year compared to baseline. Frequencies of all immune subpopulations will be calculated to identify pulmonary inflammation signatures.
6-Minute Walk Test | Baseline and one year
  Change in 6-Minute Walk Test at one year compared to baseline. The distance covered over a time of 6 minutes. Measure of cardiopulmonary exercise reserve.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Glassberg, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Mount Sinai St Luke's, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided